CLINICAL TRIAL: NCT03088033
Title: A Study to Evaluate the Corvia Medical, Inc. IASD® System II to Reduce Elevated Left Atrial Pressure in Patients With Heart Failure
Brief Title: REDUCE LAP-HF TRIAL II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1601
Record Dates: First submitted 2017-03-14; First posted 2017-03-23 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Patients randomized to the treatment arm will undergo a fluoroscopically and intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) guided trans-septal puncture and IASD System II implant procedure.
  Interventions: Device: IASD System II implant
- Control (Sham Comparator): Patients randomized to the control arm will undergo ICE from the femoral vein or TEE for examination of the atrial septum and left atrium.
  Interventions: Other: intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE)

INTERVENTIONS:
Device: IASD System II implant — The primary component of the system is an implant placed in the atrial septum designed to allow left to right flow between the left atrium and right atrium to reduce the elevated left atrial pressure.
  Arms: Treatment
Other: intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) — intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) for examination of the atrial septum and left atrium.
  Arms: Control

SUMMARY:
Multicenter, Prospective, Randomized Controlled, Blinded Trial, with a Non-implant Control group; 1:1 randomization.

DETAILED DESCRIPTION:
Following supine bicycle exercise testing to assess eligibility, the eligible patients are randomized to the treatment or control group.

All patients will be sedated, and both treatment and control arm patients will undergo placement of a femoral venous access sheath after randomization.

Patients randomized to the treatment arm will undergo a fluoroscopically and intra-cardiac echocardiography (ICE), or transesophageal echocardiography (TEE) guided trans-septal puncture and IASD System II implant procedure. Patients randomized to the control arm will undergo ICE from the femoral vein or TEE for examination of the atrial septum and left atrium.

Patients will be evaluated at pre-specified time intervals and followed for 5 years.

All patients will be unblinded after the 24 month follow up visit.

ELIGIBILITY:
SELECT INCLUSION CRITERIA

* Chronic symptomatic Heart Failure (HF) documented by one or more of the following:

  * Symptoms of HF requiring current treatment with diuretics for ≥ 30 days AND
  * NYHA class II with a history of > NYHA class II; OR NYHA class III, or ambulatory NYHA class IV symptoms (paroxysmal nocturnal dyspnea, orthopnea, dyspnea on mild or moderate exertion) at screening; or signs (any rales post cough, chest x-ray demonstrating pulmonary congestion,) within past 12 months; AND
  * ≥ 1 HF hospital admission (with HF as the primary, or secondary diagnosis); or treatment with intravenous (IV), or intensification of oral diuresis for HF in a healthcare facility within the 12 months prior to study entry; OR an NT-pro BNP value > 150 pg./ml in normal sinus rhythm, > 450 pg./ml in atrial fibrillation, or a BNP value > 50 pg./ml in normal sinus rhythm, > 150 pg./ml in atrial fibrillation within the past 6 months.
* Ongoing stable GDMT HF management and management of potential comorbidities according to the 2013 ACCF/AHA Guidelines for the management of Heart Failure (with no significant changes [>100% increase or 50% decrease], excluding diuretic dose change for a minimum of 4 weeks prior to screening) that is expected to be maintained without change for 6 months
* Age ≥ 40 years old, LV ejection fraction (EF) ≥ 40% within the past 3 months, without previously documented EF <30% (within the past 3 years)
* Elevated PCWP with a gradient compared to right atrial pressure (RAP), documented by end-expiratory PCWP during supine ergometer exercise ≥ 25mmHg, and greater than RAP by ≥ 5 mmHg

SELECT EXCLUSION CRITERIA

* MI and/or percutaneous cardiac intervention within past 3 months; CABG in past 3 months, or current indication for coronary revascularization; AVR (surgical AVR or TAVR) within the past 12 months.
* Cardiac Resynchronization Therapy initiated within the past 6 months
* Advanced heart failure defined as one or more of the below:

  * ACC/AHA/ESC Stage D heart failure, non-ambulatory NYHA Class IV HF;
  * Cardiac index < 2.0 L/min/m2
  * Inotropic infusion (continuous or intermittent) for EF< 40% within the past 6 months
  * Patient is on the cardiac transplant waiting list
* Inability to perform 6 minute walk test (distance < 50 m), OR 6 minute walk test > 600m
* History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within the past 6 months
* Presence of significant valve disease defined by the site cardiologist as:

  * Mitral valve regurgitation defined as grade ≥ 3+ MR
  * Tricuspid valve regurgitation defined as grade ≥ 2+ TR
  * Aortic valve disease defined as ≥ 2+ AR or > moderate AS
* Known clinically significant untreated carotid artery stenosis likely to require intervention
* Currently requiring dialysis; or estimated-GFR <25ml/min/1.73 m2 by CKD-Epi equation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Composite Primary Endpoint | Up to 24 months
  The primary endpoint is the composite of (a) incidence of and time-to-cardiovascular mortality or first non-fatal, ischemic stroke through 12 months; (b) total rate (first plus recurrent) per patient year of heart failure (HF) events, defined as hospital admissions, acute healthcare facility visits or urgent unscheduled outpatient visits for IV diuresis or intensification of oral diuretics for HF up to 24 months, analyzed when the last randomized subject completes 12 months follow-up, and time-to-first HF event; and (c) change in baseline KCCQ total summary score at 12 months.

SECONDARY OUTCOMES:
Composite safety endpoint defined as follows: | 12 months
  1. Cardiovascular mortality
  2. Non-fatal, ischemic stroke
  3. New onset or worsening of kidney dysfunction (defined as eGFR decrease of > 20 ml/min)
  4. Major adverse cardiac events through 12-months defined as: i. Cardiac death; ii. Myocardial infarction; iii. Cardiac tamponade; iv. Emergency cardiac surgery
  5. Thrombo-embolic complications (TIA, systemic embolization)
  6. Newly acquired persistent or permanent AF or atrial flutter through
  7. ≥30% increase in RV size/decrease in TAPSE
Rate of heart failure admissions | Up to 24 months
  Total rate (first plus recurrent) per patient year of heart failure (HF) events, defined as hospital admissions, acute healthcare facility visits, or urgent unscheduled outpatient visits for IV diuresis or intensification of oral diuretics for HF up to 24 months, analyzed when the last randomized subject completes 12-month follow-up
Change in NYHA Class | 12 months
  Change in NYHA functional Class assessed by a blinded physician between baseline and 12 months
Change in Kansas City Cardiomyopathy Questionnaire | 12 months
  Change in KCCQ score between baseline and 12 months, categorized as ≤0, >0 - 5, >5 - 10, >10 - 15, >15 - 20, >20 - 25, >25.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern Memorial Hospital; Marty Leon, MD, Principal Investigator — Columbia University
Locations (91):
- United States (44):
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - University of Arizona College of Medicine, Tucson, Arizona
  - Scripps Clinic, La Jolla, California
  - Kaiser Permanente San Diego, La Jolla, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - South Denver Cardiology Associates, Littleton, Colorado
  - Yale University, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Evanston Northshore Healthcare, Evanston, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Hackensack University Medical Center, Hamilton, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Christ Hospital Ohio Heart and Vascular Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University College of Medicine, Columbus, Ohio
  - Ohio Health, Columbus, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Australia (6):
  - Concord Hospital, Camperdown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - St. Vincent Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Medizinische Universität Graz, Graz, Austria
- Belgium (2):
  - OLVZ Aalst, Aalst
  - Az Sint-Jan Brugge, Bruges
- Hamilton Health Sciences, Hamilton, Ontario, Canada
- University Hospital Center, Zagreb, Zagreb, Croatia
- Rigshospitalet, Copenhagen, Denmark
- France (6):
  - CHU de Dijon, Dijon
  - CHU de Nantes, Nantes
  - Hôpital Bichat, Paris
  - Hôpital La Pitié Salpétrière, Paris
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
- Germany (11):
  - Kerckhoff Klinik, Bad Nauheim
  - Charite Universitatsmedizin Berlin, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Universitatklinikum Duseldorf, Düsseldorf
  - Heart Center Freiburg University, Freiburg im Breisgau
  - Georg-August-Universitat, Göttingen
  - Cardiologicum CRC, Hamburg
  - UKE Hamburg, Hamburg
  - University of Heidelberg, Heidelberg
  - Heart Center of the University of Leipzig, Leipzig
  - Klinikum der Universität Munchen, Munich
- University of Milano, Milan, Italy
- Japan (9):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kyushu University Hospital, Fukuoka
  - The Hospital of Hyogo College of Medicine, Hyōgo
  - Nara Medical University Hospital, Nara
  - National Cerebral and Cardiovascular Center, Osaka
  - Osaka University Hospital, Osaka
  - The University of Tokyo Hospital, Tokyo
  - Tottori University Hospital, Tottori
  - Toyama University Hospital, Toyama
- Netherlands (4):
  - VU University Medical Center, Amsterdam
  - UMC Groningen, Groningen
  - Maastricht UMC Hart & Vaat Centrum, Maastricht
  - St Antonius Ziekenhuis, Nieuwegein
- Fourth Military Hospital, Wroclaw, Poland
- Hospital Clinic Barcelona, Barcelona, Spain
- United Kingdom (2):
  - Golden Jubilee Hospital, Glasgow
  - Guys & St Thomas NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaudhary RS, Hussain SMD, Wang YS, Komtebedde J, Hasenfuss G, Borlaug BA, Kaye DM, Cleland JGF, Leon MB, Shah SJ, van Veldhuisen DJ, Solomon SD, Cikes M, Cutlip DE. Expanded Definition of Worsening Heart Failure: Impact on Clinical Outcomes and Quality-of-Life Assessment. JACC Heart Fail. 2025 Sep;13(9):102571. doi: 10.1016/j.jchf.2025.102571. Epub 2025 Jul 25. PMID 40714684
- [Derived] Litwin SE, Komtebedde J, Borlaug BA, Kaye DM, Hasenfubeta G, Kawash R, Hoendermis E, Hummel SL, Cikes M, Gustafsson F, Chung ES, Mohan RC, Sverdlov AL, Swarup V, Winkler S, Hayward CS, Bergmann MW, Bugger H, McKenzie S, Nair A, Rieth A, Burkhoff D, Cutlip DE, Solomon SD, van Veldhuisen DJ, Leon MB, Shah SJ. Long term safety and outcomes after atrial shunting for heart failure with preserved or mildly reduced ejection fraction: 5-year and 3-year follow-up in the REDUCE LAP-HF I and II trials. Am Heart J. 2024 Dec;278:106-116. doi: 10.1016/j.ahj.2024.08.014. Epub 2024 Sep 3. PMID 39237070
- [Derived] Gustafsson F, Petrie MC, Komtebedde J, Swarup V, Winkler S, Hasenfuss G, Borlaug BA, Mohan RC, Flaherty JD, Sverdlov AL, Fail PS, Chung ES, Lurz P, Lilly S, Kaye DM, Cleland JGF, Cikes M, Leon MB, Cutlip DE, van Veldhuisen DJ, Solomon SD, Shah SJ. 2-Year Outcomes of an Atrial Shunt Device in HFpEF/HFmrEF: Results From REDUCE LAP-HF II. JACC Heart Fail. 2024 Aug;12(8):1425-1438. doi: 10.1016/j.jchf.2024.04.011. Epub 2024 Jun 26. PMID 38934964
- [Derived] Patel RB, Silvestry FE, Komtebedde J, Solomon SD, Hasenfuss G, Litwin SE, Borlaug BA, Price MJ, Kawash R, Hummel SL, Cutlip DE, Leon MB, van Veldhuisen DJ, Rieth AJ, McKenzie S, Bugger H, Mazurek JA, Kapadia SR, Vanderheyden M, Ky B, Shah SJ. Atrial Shunt Device Effects on Cardiac Structure and Function in Heart Failure With Preserved Ejection Fraction: The REDUCE LAP-HF II Randomized Clinical Trial. JAMA Cardiol. 2024 Jun 1;9(6):507-522. doi: 10.1001/jamacardio.2024.0520. PMID 38630494
- [Derived] Patel RB, Reddy VY, Komtebedde J, Wegerich SW, Sekaric J, Swarup V, Walton A, Laurent G, Chetcuti S, Rademann M, Bergmann M, McKenzie S, Bugger H, Bruno RR, Herrmann HC, Nair A, Gupta DK, Lim S, Kapadia S, Gordon R, Vanderheyden M, Noel T, Bailey S, Gertz ZM, Trochu JN, Cutlip DE, Leon MB, Solomon SD, van Veldhuisen DJ, Auricchio A, Shah SJ. Atrial Fibrillation Burden and Atrial Shunt Therapy in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2023 Oct;11(10):1351-1362. doi: 10.1016/j.jchf.2023.05.024. Epub 2023 Jul 19. PMID 37480877
- [Derived] Litwin SE, Komtebedde J, Hu M, Burkhoff D, Hasenfuss G, Borlaug BA, Solomon SD, Zile MR, Mohan RC, Khawash R, Sverdlov AL, Fail P, Chung ES, Kaye DM, Blair J, Eicher JC, Hummel SL, Zirlik A, Westenfeld R, Hayward C, Gorter TM, Demers C, Shetty R, Lewis G, Starling RC, Patel S, Gupta DK, Morsli H, Penicka M, Cikes M, Gustafsson F, Silvestry FE, Rowin EJ, Cutlip DE, Leon MB, Kitzman DW, Kleber FX, Shah SJ; REDUCE LAP-HF Investigators and Research Staff. Exercise-Induced Left Atrial Hypertension in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2023 Aug;11(8 Pt 2):1103-1117. doi: 10.1016/j.jchf.2023.01.030. Epub 2023 Mar 20. PMID 36939661
- [Derived] Shah SJ, Borlaug BA, Chung ES, Cutlip DE, Debonnaire P, Fail PS, Gao Q, Hasenfuss G, Kahwash R, Kaye DM, Litwin SE, Lurz P, Massaro JM, Mohan RC, Ricciardi MJ, Solomon SD, Sverdlov AL, Swarup V, van Veldhuisen DJ, Winkler S, Leon MB; REDUCE LAP-HF II investigators. Atrial shunt device for heart failure with preserved and mildly reduced ejection fraction (REDUCE LAP-HF II): a randomised, multicentre, blinded, sham-controlled trial. Lancet. 2022 Mar 19;399(10330):1130-1140. doi: 10.1016/S0140-6736(22)00016-2. Epub 2022 Feb 1. PMID 35120593